CLINICAL TRIAL: NCT01541098
Title: A Phase II Clinical Study of Lyophilized Plasma in Patients on Warfarin
Brief Title: A Clinical Study of Lyophilized Plasma in Patients on Warfarin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2011-I-LyP-1
Record Dates: First submitted 2012-02-16; First posted 2012-02-29 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Anticoagulant Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Licensed Plasma (Active Comparator)
  Interventions: Biological: Licensed Plasma
- Lyophilized Plasma (Experimental)
  Interventions: Biological: Lyophilized Plasma

INTERVENTIONS:
Biological: Lyophilized Plasma — Licensed plasma that has been lyophilized.
  Arms: Lyophilized Plasma
Biological: Licensed Plasma — Plasma that has been authorized for transfusion.
  Arms: Licensed Plasma

SUMMARY:
This is a multi center, phase 2 randomized controlled study to determine the effect of lyophilized plasma in patients on warfarin therapy.

ELIGIBILITY:
Inclusion Criteria

1. Patients receiving oral anticoagulation with warfarin derived agents.
2. Patients who have need for urgent surgery, an invasive procedure or identification of a patient with active bleeding where oral or parenteral vitamin K therapy is deemed too slow in its action for reversal of warfarin anticoagulant effects.
3. Patients with an elevated international normalized ratio.

Exclusion Criteria

1. Patients who are clinically unstable.
2. Patients who have congenital or acquired coagulopathies (other than warfarin therapy).
3. Patients who have received medications that could interfere with the results of laboratory testing.
4. Pregnant or nursing women.
5. Patients participating in another clinical treatment study currently or during the past 1 month prior to study inclusion.
6. Patients previously enrolled in this study.
7. Active illicit drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Assess and Compare Adverse Events | Duration of Study (Less than or equal to 72 hours)
  The primary safety objective is to assess the adverse events after infusion of lyophilized plasma compared to control.